CLINICAL TRIAL: NCT01227629
Title: Dose Exploration in Patients With Atrial Fibrillation
Brief Title: PETRO Stroke Prevention in Patients With AF by Treatment With Dabigatran, With and Without Aspirin, Compared to Warfarin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 1160.20; PETRO trial (Other: OTHER)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Warfarin

ARMS (10):
- dabigatran 50 mg twice daily (bid) (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. Twice daily (bis in die = bid).
  Interventions: Drug: dabigatran without ASA
- dabigatran 50 mg bid + 81 mg ASA qd (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. Acetylsalicylic acid (ASA) once daily (quaque dies = qd) in the morning.
  Interventions: Drug: dabigatran with ASA
- dabigatran 50 mg bid + 325 mg ASA qd (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. ASA in the morning
  Interventions: Drug: dabigatran with ASA
- dabigatran 150 mg bid (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening
  Interventions: Drug: dabigatran without ASA
- dabigatran 150 mg bid + 81 mg ASA qd (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. ASA in the morning
  Interventions: Drug: dabigatran with ASA
- dabigatran 150 mg bid + 325 mg ASA qd (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. ASA in the morning
  Interventions: Drug: dabigatran with ASA
- dabigatran 300 mg bid (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening
  Interventions: Drug: dabigatran without ASA
- dabigatran 300 mg bid + 81 mg ASA qd (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. ASA in the morning
  Interventions: Drug: dabigatran with ASA
- dabigatran 300 mg bid + 325 mg ASA qd (Experimental): Dabigatran: one capsule in the morning and 1 capsule in the evening. ASA in the morning
  Interventions: Drug: dabigatran with ASA
- warfarin (Active Comparator): once daily, dosed to target International Normalised Ratio (INR) 2.0 to 3.0
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: dabigatran with ASA — dose comparison in combination
  Arms: dabigatran 50 mg bid + 81 mg ASA qd
Drug: dabigatran with ASA — dose comparison in combination
  Arms: dabigatran 50 mg bid + 325 mg ASA qd
Drug: dabigatran with ASA — dose comparison in combination
  Arms: dabigatran 150 mg bid + 81 mg ASA qd
Drug: dabigatran with ASA — dose comparison in combination
  Arms: dabigatran 150 mg bid + 325 mg ASA qd
Drug: dabigatran with ASA — dose comparison in combination
  Arms: dabigatran 300 mg bid + 81 mg ASA qd
Drug: dabigatran with ASA — dose comparison in combination
  Arms: dabigatran 300 mg bid + 325 mg ASA qd
Drug: warfarin — comparator
  Arms: warfarin
Drug: dabigatran without ASA — dose comparison
  Arms: dabigatran 50 mg twice daily (bid)
Drug: dabigatran without ASA — dose comparison
  Arms: dabigatran 150 mg bid
Drug: dabigatran without ASA — dose comparison
  Arms: dabigatran 300 mg bid

SUMMARY:
The purpose of this trial is to evaluate the safety of different doses of BIBR 1048, alone or in combination with acetylsalicylic acid (ASA), as determined by the rates of bleeding and other adverse events.

A secondary objective of this trial is to evaluate the anticoagulant effect of different doses of BIBR 1048, based on the reduction of plasma concentrations of D-dimer, a laboratory marker for activated coagulation in patients with atrial fibrillation (AF), and to correlate bleeding and other events with pharmacokinetic (PK) and pharmacodynamic (PD) data.

ELIGIBILITY:
Inclusion criteria

1. Non-rheumatic atrial fibrillation.
2. Coronary artery disease (CAD), documented by previous myocard infarction (MI), angina, positive stress test, previous coronary intervention or bypass surgery, or atherosclerotic lesion(s) diagnosed by coronary angiography) is only considered as one of several possible qualifying risk factors. After recruitment of ca. 30%, a protocol amendment 4 was issued so that CAD was only considered as one of several possible qualifying risk factors, 2. see (3 f) below.
3. An additional risk factor for stroke, i.e. one or more of the following conditions/events:

   1. hypertension (defined as systolic bloodpressure (SBP) > 140 mmHg and/or diastolic bloodpressure (DBP) > 90 mm Hg) requiring antihypertensive medical treatment.
   2. diabetes mellitus (type I and II).
   3. symptomatic heart failure or left ventricular dysfunction (ejection fraction (EF) < 40%).
   4. a previous ischemic stroke or transient ischemic attack.
   5. age greater than 75 years.
   6. history of coronary artery disease (by amendment 4)
4. Treatment with warfarin or other vitamin K dependent anticoagulants for at least 8 weeks prior to inclusion. International normalised ratio (INR) should be within therapeutic range (i.e. INR 2.0 - 3.0) at visit 1 otherwise the visit should be rescheduled.
5. Age > = 18 years at entry.
6. Written, informed consent.

Exclusion criteria

1. Valvular heart disease.
2. Planned cardioversion.
3. Recent (=< 1 month) myocardial infarction, stroke or transient ischemic attack (TIA), or patients who have received a coronary stent within the last 6 months.
4. Intolerance or contraindications to acetylsalicylic acid (ASA).
5. Any contraindication to anticoagulant therapy.
6. Major bleeding within the last 6 months (other than gastrointestinal (GI) hemorrhage).
7. Severe renal impairment (estimated glomerular filtration rate (GFR) =< 30 mL/min).
8. Uncontrolled hypertension (SBP > 180 mmHg and/or DBP > 100 mmHg).
9. Abnormal liver function as defined by aspartat-aminotransferase (AST), alanin-aminotransferase (ALT), serum bilirubin or alkaline phosphatase (AP) above the reference range, or history of liver disease.
10. Women who are pregnant or of childbearing potential who refuses to use a medically acceptable form of contraception throughout the study.
11. Patients who have received an investigational drug within the last 30 days.
12. Patients scheduled for major surgery or invasive procedures which may cause bleeding, or those who have had major surgery or percutaneous coronary intervention (PCI) within 6 weeks.
13. Patients considered unreliable by the investigator.
14. Another indication for anticoagulant treatment.
15. Patients suffering from anemia.
16. Patients suffering from thrombocytopenia.
17. Any other condition which, in the discretion of the investigator, would not allow safe participation in the study.
18. Concomitant treatment with antiplatelet agents other than ASA.
19. Recent malignancy or radiation therapy (=< 6 month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2003-09; Primary Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (38):
- United States (14):
  - 1160.20.10010, Fayetteville, Arkansas
  - 1160.20.10003 La Mesa Cardiac, La Mesa, California
  - 1160.20.10006 The Ford Research Institute, PA, Pensacola, Florida
  - 1160.20.10004, Port Charlotte, Florida
  - 1160.20.10002, St. Petersburg, Florida
  - 1160.20.10015, Baltimore, Maryland
  - 1160.20.10008, Westminister, Maryland
  - 1160.20.10012, Pittsfield, Massachusetts
  - 1160.20.10007, Troy, Michigan
  - 1160.20.10014, Hawthorne, New York
  - 1160.20.10013, New Hyde Park, New York
  - 1160.20.10009, North Durham, North Carolina
  - 1160.20.10001, Philadelphia, Pennsylvania
  - 1160.20.10005, Germantown, Tennessee
- Denmark (13):
  - 1160.20.45010, Aalborg
  - 1160.20.45005 Aarhus Sygehus, Aarhus C
  - 1160.20.45007 Medicinsk afdeling, Brædstrup
  - 1160.20.45003 Forskningscentret plan 3, Elsinore
  - 1160.20.45011 Medicinsk afd., Esbjerg
  - 1160.20.45012 Afdeling B3, Frederikssund
  - 1160.20.45004 Herlev Hospital, Herlev
  - 1160.20.45009 Medicinsk amb. B8, Holbæk
  - 1160.20.45002 Kardiologisk afdeling, Hvidovre
  - 1160.20.45014 Hjertemedicinsk afd., Køge
  - 1160.20.45001 Kardiologisk Laboratorium, Odense
  - 1160.20.45013 Kardiologisk afd., Roskilde
  - 1160.20.45006 Medicinsk afdeling, Svendborg
- Sweden (11):
  - 1160.20.46013 HIA, Mälarsjukhuset, Eskilstuna
  - 1160.20.46007 Falu Lasarett, Falun
  - 1160.20.46005 Ryhovs Länssjukhus, Jönköping
  - 1160.20.46010 Länssjukhuset Kalmar, Kalmar
  - 1160.20.46009 Universitetssjukhuset MAS, Malmo
  - 1160.20.46008 Vrinnevisjukhuset, Norrköping
  - 1160.20.46004 Universitetssjukhuset, Örebro
  - 1160.20.46002 Södersjukhuset, Stockholm
  - 1160.20.46011 Arytmienheten, Med klin, Stockholm
  - 1160.20.46006 Norrlands Universitetssjukhus, Umeå
  - 1160.20.46003 Centrallasarettet, Västerås

RESULTS

PARTICIPANT FLOW:
Groups:
- BIBR 1048 50 mg b.i.d; BIBR 1048 150 mg b.i.d; BIBR 1048 300 mg b.i.d: bid (twice daily) oral
- BIBR 1048 50 mg b.i.d + ASA 81 mg q.d.; BIBR 1048 50 mg b.i.d + ASA 325 mg qd; BIBR 1048 150 mg b.i.d + ASA 81 mg qd; BIBR 1048 150 mg b.i.d + ASA 325 mg qd; BIBR 1048 300 mg b.i.d + ASA 81 mg qd; BIBR 1048 300 mg b.i.d + ASA 325 mg qd: bid (twice daily) oral + qd (once daily) oral
- Warfarin, Dosed to Target INR 2.0 to 3.0: qd (once daily) oral
Period: Overall Study
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Started | 58 (Started: Participant was randomised and took at least one dose of randomised study medication) | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Completed | 56 (Completed: Participant without premature discontinuation in the randomised treatment period) | 18 | 26 | 91 | 32 | 32 | 90 | 27 | 24 | 68
Not Completed | 2 | 2 | 1 | 8 | 2 | 1 | 8 | 6 | 6 | 2
Not completed — Adverse Event | 2 | 2 | 1 | 6 | 1 | 1 | 6 | 6 | 4 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0 | Total
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70 | 502
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (8.8) | 70.1 (9.4) | 71.6 (8.1) | 69.7 (7.7) | 72.1 (9.0) | 69.7 (8.0) | 69.0 (9.1) | 71.8 (7.2) | 68.6 (7.1) | 69.0 (8.3) | 69.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 5 | 15 | 8 | 8 | 19 | 7 | 2 | 11 | 91
  Male | 46 | 16 | 22 | 84 | 26 | 25 | 79 | 26 | 28 | 59 | 411
Baseline documentation regarding the atrial fibrillation [Number; unit: Participants]
  Persistent | 20 | 9 | 10 | 43 | 13 | 10 | 37 | 14 | 12 | 27 | 195
  Permanent | 23 | 9 | 11 | 35 | 11 | 16 | 37 | 10 | 14 | 26 | 192
  Paroxysmal | 15 | 2 | 6 | 21 | 10 | 7 | 24 | 9 | 4 | 17 | 115
Baseline documentation regarding stroke [Number; unit: Participants] — Documentation of stroke as specific risk factor
  Participants
    No | 54 | 18 | 24 | 93 | 30 | 30 | 91 | 31 | 26 | 62 | 459
    Yes | 4 | 2 | 3 | 6 | 4 | 3 | 7 | 2 | 4 | 8 | 43
Baseline documentation regarding transient ischemic attack [Number; unit: Participants] — Documentation of transient ischemic attack as specific risk factor
  Participants
    No | 49 | 20 | 25 | 88 | 31 | 31 | 90 | 30 | 26 | 63 | 453
    Yes | 9 | 0 | 2 | 11 | 3 | 2 | 8 | 3 | 4 | 7 | 49
Baseline documentation regarding transient ischemic attack or stroke [Number; unit: Participants] — Documentation of transient ischemic attack or stroke as specific risk factor
  Participants
    No | 45 | 18 | 23 | 82 | 27 | 28 | 85 | 28 | 22 | 57 | 415
    Yes | 13 | 2 | 4 | 17 | 7 | 5 | 13 | 5 | 8 | 13 | 87
Baseline documentation regarding hypertension [Number; unit: Participants] — Documentation of hypertension as specific risk factor
  Participants
    No | 17 | 10 | 8 | 21 | 13 | 14 | 24 | 8 | 10 | 21 | 146
    Yes | 41 | 10 | 19 | 78 | 21 | 19 | 74 | 25 | 20 | 49 | 356
Baseline documentation regarding symptomatic heart failure [Number; unit: Participants] — Documentation of symptomatic heart failure as specific risk factor
  Participants
    No | 41 | 12 | 17 | 73 | 20 | 21 | 85 | 20 | 20 | 46 | 355
    Yes | 17 | 8 | 10 | 26 | 14 | 12 | 13 | 13 | 10 | 24 | 147
Baseline documentation regarding left ventricular dysfunction [Number; unit: Participants] — Documentation of left ventricular dysfunction as specific risk factor
  Participants
    No | 41 | 14 | 17 | 68 | 22 | 19 | 78 | 20 | 14 | 44 | 337
    Yes | 17 | 6 | 10 | 31 | 12 | 14 | 20 | 13 | 16 | 26 | 165
Baseline documentation regarding symptomatic heart failure or left ventricular dysfunction [Number; unit: Participants] — Documentation of symptomatic heart failure or left ventricular dysfunction as specific risk factor
  Participants
    No | 35 | 10 | 14 | 55 | 15 | 17 | 71 | 14 | 12 | 34 | 277
    Yes | 23 | 10 | 13 | 44 | 19 | 16 | 27 | 19 | 18 | 36 | 225
Coronary Artery Disease [Number; unit: participants] — Documentation of Coronary Artery Disease as inclusion criterion or specific risk factor
  participants
    no | 39 | 1 | 1 | 55 | 3 | 4 | 62 | 2 | 1 | 28 | 196
    yes | 19 | 19 | 26 | 44 | 31 | 29 | 36 | 31 | 29 | 42 | 306
D-dimer at baseline N=(56;19;25;88;29;32;85;31;29;63;457) [Mean (Standard Deviation); unit: ng/ml] | 106.8 (104.1) | 104.5 (62.9) | 176.9 (389.9) | 100.8 (94.5) | 120.3 (95.4) | 96.3 (64.3) | 146.8 (210.9) | 119.4 (95.5) | 83.8 (48.8) | 139.9 (251.9) | 120.9 (173.7)
Soluble fibrin at baseline N=(53;16;23;88;27;29;92;30;25;65;448) [Mean (Standard Deviation); unit: µg/ml] | 4.9 (4.4) | 5.3 (7.9) | 5.4 (5.9) | 5.8 (8.8) | 9.1 (15.5) | 7.6 (14.8) | 7.4 (11.5) | 9.2 (26.0) | 6.5 (9.2) | 7.2 (10.4) | 6.8 (11.9)
Thromboxane B2 (TXB2) measured at baseline N=(53;20;23;93;30;30;90;31;30;67;467) [Mean (Standard Deviation); unit: pg/mg Creatinine] | 3968.5 (2530.4) | 3795.9 (2252.9) | 4705.6 (3047.5) | 4138.1 (2184.6) | 4485.7 (2147.8) | 4084.9 (2253.5) | 3619.0 (2020.6) | 4450.8 (2653.7) | 3735.6 (2440.6) | 4177.9 (2661.2) | 4051.6 (2367.7)
ECT at baseline N=(57;20;27;98;34;33;95;33;29;56;482) [Mean (Standard Deviation); unit: seconds] | 32.3 (2.0) | 31.8 (1.9) | 31.9 (2.2) | 31.9 (2.2) | 32.0 (1.9) | 32.6 (2.4) | 33.6 (13.3) | 31.9 (1.8) | 32.2 (2.6) | 32.0 (2.4) | 32.4 (6.2)
aPTT at baseline N=(57;20;27;98;34;33;96;33;29;57;484) [Mean (Standard Deviation); unit: seconds] | 32.5 (3.0) | 31.2 (3.5) | 32.4 (3.6) | 34.2 (15.2) | 33.5 (7.6) | 34.2 (6.7) | 32.8 (5.7) | 32.6 (3.4) | 32.9 (6.7) | 33.2 (3.7) | 33.1 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fatal or Life-threatening Major Bleeding Events
Description: Retroperitoneal, intracranial, intraocular, or intraspinal bleeding, or requiring surgical treatment, or leading to a transfusion of 2 units or more, or leading to a fall in hemoglobin of 20g/L or more
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 59 | 21 | 27 | 100 | 36 | 33 | 105 | 34 | 30 | 70
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0

2. Primary Outcome: Number of Participants With Minor/Relevant Bleeding Events
Description: Haematuria, rectal bleeding, gingival bleeding, skin hematoma of 25cm^2 or more, nose bleed of more than 5 minutes duration, bleeding leading to a hospitalization, leading to a transfusion of less than 2 units or any other clinically relevant bleeding
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons were performed, due to the small number of events per group
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 59 | 21 | 27 | 100 | 36 | 33 | 105 | 34 | 30 | 70
Participants | 0 | 1 | 1 | 9 | 2 | 2 | 6 | 4 | 3 | 4

3. Primary Outcome: Number of Participants With Minor/Nuisance Bleeding Events
Description: All bleeding events not fulfilling one of the criteria for major bleeding event or minor/relevant bleeding events.
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons were performed, due to the small number of events per group
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 59 | 21 | 27 | 100 | 36 | 33 | 105 | 34 | 30 | 70
Participants | 2 | 1 | 2 | 6 | 6 | 5 | 9 | 7 | 9 | 9

4. Secondary Outcome: Number of Participants With Thromboembolic Events: Composite Endpoint
Description: Combination of ischemic stroke (fatal or non fatal), transient ischemic attack, systemic thromboembolism, myocardial infarction (fatal or non fatal), other major adverse cardiac event and all cause mortality
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Thromboembolic Events: Ischemic Stroke
Description: Occurence of an ischemic stroke (fatal or non-fatal)
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants
  None | 58 | 19 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
  Fatal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-Fatal | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Both | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Thromboembolic Events: Number of Participants With Transient Ischemic Attack
Description: Occurence of a transient ischemic attack
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Thromboembolic Events: Number of Participants With Systemic Thromboembolism
Description: Occurence of a systemic thromboembolism
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Thromboembolic Events: Number of Participants With Myocardial Infarction
Description: Occurence of a myocardial infarction
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants
  None | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
  Fatal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-Fatal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Both | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Thromboembolic Events: Number of Participants With Other Major Cardiac Events
Description: Occurence of other major adverse cardiac events
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Thromboembolic Events: Number of Participants Who Died
Description: Occurence of death by all causes
Time Frame: 12 weeks
Population: All randomized patients. No statistical comparisons were performed, due to the extremely small number of events.
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: D-dimer: Difference From Baseline
Description: Difference in D-dimer from baseline to last available value
Time Frame: baseline and 12 weeks
Population: All randomised patients, only per-protocol data included.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 55 | 19 | 26 | 87 | 29 | 32 | 88 | 29 | 29 | 63
ng/ml | 22.3 (65.4) | 12.3 (25.3) | 50.2 (182.8) | 8.1 (41.6) | 29.1 (90.4) | 8.6 (49.2) | 4.2 (95.8) | 11.3 (82.2) | -7.9 (40.9) | -5.8 (50.6)
Statistical Analysis 1: Comparison: BIBR 1048 50 mg b.i.d vs BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. vs BIBR 1048 50 mg b.i.d + ASA 325 mg qd vs BIBR 1048 150 mg b.i.d vs BIBR 1048 150 mg b.i.d + ASA 81 mg qd vs BIBR 1048 150 mg b.i.d + ASA 325 mg qd vs BIBR 1048 300 mg b.i.d vs BIBR 1048 300 mg b.i.d + ASA 81 mg qd vs BIBR 1048 300 mg b.i.d + ASA 325 mg qd vs Warfarin, Dosed to Target INR 2.0 to 3.0; Group comparison of differences from baseline to last available value; Test type: Superiority or Other; p = 0.0357, Kruskal-Wallis

12. Secondary Outcome: Soluble Fibrin: Difference From Baseline
Description: Difference from baseline to visit 7
Time Frame: baseline and 12 weeks
Population: All randomised patients, only per-protocol data included.
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 52 | 15 | 25 | 88 | 25 | 24 | 83 | 27 | 20 | 54
µg/ml | 3.2 (22.0) | 0.9 (2.3) | 1.2 (8.4) | 0.3 (5.1) | -2.0 (9.9) | -1.3 (8.8) | 2.3 (26.8) | -0.7 (4.6) | -1.9 (12.0) | 0.1 (4.0)
Statistical Analysis 1: Comparison: BIBR 1048 50 mg b.i.d vs BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. vs BIBR 1048 50 mg b.i.d + ASA 325 mg qd vs BIBR 1048 150 mg b.i.d vs BIBR 1048 150 mg b.i.d + ASA 81 mg qd vs BIBR 1048 150 mg b.i.d + ASA 325 mg qd vs BIBR 1048 300 mg b.i.d vs BIBR 1048 300 mg b.i.d + ASA 81 mg qd vs BIBR 1048 300 mg b.i.d + ASA 325 mg qd vs Warfarin, Dosed to Target INR 2.0 to 3.0; Group comparison of differences from baseline to week 12; Test type: Superiority or Other; p = 0.26711, Kruskal-Wallis

13. Secondary Outcome: 11-dehydrothromboxane B2 (TXB2): Difference From Baseline
Description: Difference from baseline to visit 7
Time Frame: baseline and 12 weeks
Population: All treated patients. No statistical comparisons due to high variability
Measure: Mean (Standard Deviation); unit: pg/mg Creatinine
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 44 | 17 | 19 | 73 | 25 | 27 | 73 | 25 | 25 | 51
pg/mg Creatinine | 596.5 (2896.3) | -1816.8 (2186.1) | -2779.8 (2953.3) | 922.0 (3874.0) | -1988.6 (2187.5) | -1125.9 (3566.6) | 1059.7 (2216.8) | -1822.6 (2381.7) | -1337.8 (2279.2) | 203.5 (2109.0)

14. Secondary Outcome: Ecarin Clotting Time (ECT): Difference From Baseline
Time Frame: baseline and 12 weeks
Population: All treated patients. No statistical comparisons due to high variability
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 56 | 19 | 26 | 94 | 34 | 33 | 86 | 29 | 27 | 27
seconds | 9.7 (8.2) | 12.0 (10.7) | 12.0 (9.6) | 31.9 (26.2) | 42.5 (29.2) | 32.7 (23.1) | 63.6 (44.8) | 70.8 (60.3) | 74.0 (70.5) | 3.1 (2.5)

15. Secondary Outcome: Activated Partial Thromboplastin Time (aPTT): Difference From Baseline
Time Frame: baseline and 12 weeks
Population: All treated patients. No statistical comparisons due to high variability
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 56 | 19 | 26 | 92 | 33 | 33 | 87 | 29 | 27 | 27
seconds | 6.4 (5.6) | 8.3 (6.1) | 8.8 (9.4) | 13.5 (18.3) | 24.9 (26.1) | 14.5 (11.5) | 25.0 (12.4) | 23.4 (12.7) | 27.2 (24.2) | 8.8 (6.7)

16. Secondary Outcome: Trough Plasma Concentration of Dabigatran (BIBR 953)
Description: The values of the trough plasma concentration of dabigatran (BIBR 953) are the by-patient geometric means of week 1, 4 and 12.
Time Frame: 12 weeks
Population: All treated patients
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 97 | 33 | 30 | 70
ng/ml | 29.1 (16.6) | 30.4 (16.6) | 31.8 (20.0) | 82.8 (54.3) | 103.2 (69.0) | 90.1 (52.5) | 188.0 (117.3) | 203.7 (123.9) | 207.6 (108.7) | NA (NA)

17. Secondary Outcome: Number of Participants With Increase of Aspartat-Aminotransferase (AST) to >2*Baseline
Description: Increase of AST to more than two times the baseline value
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons due to extremely small number of cases
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  No | 57 | 20 | 24 | 93 | 32 | 31 | 95 | 31 | 30 | 68
  Yes | 1 | 0 | 3 | 6 | 2 | 2 | 2 | 1 | 0 | 1

18. Secondary Outcome: Number of Participants With Increase of Alkaline Phosphatase (AP) to >2*Baseline
Description: Increase of AP to more than two times the baseline value
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons due to extremely small number of cases
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  No | 58 | 20 | 27 | 98 | 33 | 33 | 97 | 32 | 29 | 69
  Yes | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0

19. Secondary Outcome: Number of Participants With Increase of Bilirubin to >2*Baseline
Description: Increase of Bilirubin to more than two times the baseline value
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons due to extremely small number of cases
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  No | 55 | 18 | 25 | 86 | 31 | 33 | 88 | 29 | 29 | 63
  Yes | 3 | 2 | 2 | 13 | 3 | 0 | 9 | 3 | 1 | 6

20. Secondary Outcome: Number of Participants With Increase of Alanine-Aminotransferase (ALT) to >2*Baseline
Description: Number of Participants with Increase of ALT to more than two times the baseline value
Time Frame: 12 weeks
Population: All treated patients. No statistical comparisons due to extremely small number of cases
Measure: Number; unit: Participants
Arm/Group | BIBR 1048 50 mg b.i.d | BIBR 1048 50 mg b.i.d + ASA 81 mg q.d. | BIBR 1048 50 mg b.i.d + ASA 325 mg qd | BIBR 1048 150 mg b.i.d | BIBR 1048 150 mg b.i.d + ASA 81 mg qd | BIBR 1048 150 mg b.i.d + ASA 325 mg qd | BIBR 1048 300 mg b.i.d | BIBR 1048 300 mg b.i.d + ASA 81 mg qd | BIBR 1048 300 mg b.i.d + ASA 325 mg qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 58 | 20 | 27 | 99 | 34 | 33 | 98 | 33 | 30 | 70
Participants
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  No | 55 | 18 | 26 | 95 | 33 | 32 | 93 | 31 | 30 | 64
  Yes | 3 | 2 | 1 | 4 | 1 | 1 | 4 | 1 | 0 | 5

21. Secondary Outcome: Severity of Adverse Events
Description: Total number of patients with any adverse event of worst intensity 'mild', 'moderate' and 'severe'.
Time Frame: 12 weeks
Population: Treated patients(Numbers of patients for adverse events are counted for each treatment and are in their sum greater than the total number of patients randomized as 14 patients on Dabigatran with ASA changed treatment,12 patients down titrated Dabigatran bid to qd of which one did the down titration at the same time as the stop of the ASA treatment)
Measure: Number; unit: participants
Groups:
- D50bid: Dabigatran 50 mg twice daily
- D50qd: Dabigatran 50 mg once daily
- D50bid + ASA81qd: Dabigatran 50 mg twice daily + ASA 81 mg once daily
- D50bid + ASA325qd: Dabigatran 50 mg twice daily + ASA 325 mg once daily
- D150bid: Dabigatran 150 mg twice daily
- D150qd: Dabigatran 150 mg once daily
- D150bid + ASA81qd: Dabigatran 150 mg twice daily + ASA 81 mg once daily
- D150qd + ASA81qd: Dabigatran 150 mg once daily + ASA 81 mg once daily
- D150bid + ASA325qd: Dabigatran 150 mg twice daily + ASA 325 mg once daily
- D150qd + ASA325qd: Dabigatran 150 mg once daily + ASA 325 mg once daily
- D300bid: Dabigatran 300 mg twice daily
- D300qd: Dabigatran 300 mg once daily
- D300bid + ASA81qd: Dabigatran 300 mg twice daily + ASA 81 mg once daily
- D300qd + ASA81qd: Dabigatran 300 mg once daily + ASA 81 mg once daily
- D300bid + ASA325qd: Dabigatran 300 mg twice daily + ASA 325 mg once daily
- D300qd + ASA325qd: Dabigatran 300 mg once daily + ASA 325 mg once daily
- Warfarin, Dosed to Target INR 2.0 to 3.0: Warfarin once daily
Arm/Group | D50bid | D50qd | D50bid + ASA81qd | D50bid + ASA325qd | D150bid | D150qd | D150bid + ASA81qd | D150qd + ASA81qd | D150bid + ASA325qd | D150qd + ASA325qd | D300bid | D300qd | D300bid + ASA81qd | D300qd + ASA81qd | D300bid + ASA325qd | D300qd + ASA325qd | Warfarin, Dosed to Target INR 2.0 to 3.0
Number analyzed (Participants) | 59 | 1 | 21 | 27 | 100 | 3 | 36 | 1 | 33 | 1 | 105 | 3 | 34 | 2 | 30 | 1 | 70
participants
  Mild | 24 | 0 | 9 | 16 | 54 | 1 | 23 | 0 | 17 | 0 | 47 | 1 | 23 | 2 | 23 | 1 | 30
  Moderate | 13 | 0 | 6 | 7 | 19 | 0 | 9 | 0 | 4 | 0 | 23 | 0 | 5 | 1 | 11 | 1 | 14
  Severe | 3 | 0 | 1 | 1 | 4 | 0 | 2 | 0 | 1 | 0 | 6 | 0 | 1 | 0 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Note that it was foreseen per protocol that all treatments were possibly to be down-titrated to BIBR 1048 q.d.; criteria included creatinine clearance and aPTT. Events are counted to the treatment on which they occurred.
Groups:
- Warfarin: Warfarin once daily
Arm/Group | D50bid | D50qd | D50bid + ASA81qd | D50bid + ASA325qd | D150bid | D150qd | D150bid + ASA81qd | D150qd + ASA81qd | D150bid + ASA325qd | D150qd + ASA325qd | D300bid | D300qd | D300bid + ASA81qd | D300qd + ASA81qd | D300bid + ASA325qd | D300qd + ASA325qd | Warfarin
Serious Adverse Events (participants affected / at risk) | 5/59 | 0/1 | 2/21 | 1/27 | 10/100 | 0/3 | 4/36 | 0/1 | 2/33 | 0/1 | 3/105 | 0/3 | 4/34 | 0/2 | 4/30 | 0/1 | 2/70
Other Adverse Events (participants affected / at risk) | 20/59 | 0/1 | 9/21 | 14/27 | 43/100 | 1/3 | 19/36 | 0/1 | 15/33 | 0/1 | 35/105 | 1/3 | 20/34 | 2/2 | 18/30 | 1/1 | 22/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D50bid (N=59) | D50qd (N=1) | D50bid + ASA81qd (N=21) | D50bid + ASA325qd (N=27) | D150bid (N=100) | D150qd (N=3) | D150bid + ASA81qd (N=36) | D150qd + ASA81qd (N=1) | D150bid + ASA325qd (N=33) | D150qd + ASA325qd (N=1) | D300bid (N=105) | D300qd (N=3) | D300bid + ASA81qd (N=34) | D300qd + ASA81qd (N=2) | D300bid + ASA325qd (N=30) | D300qd + ASA325qd (N=1) | Warfarin (N=70)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic inspiratory decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D50bid (N=59) | D50qd (N=1) | D50bid + ASA81qd (N=21) | D50bid + ASA325qd (N=27) | D150bid (N=100) | D150qd (N=3) | D150bid + ASA81qd (N=36) | D150qd + ASA81qd (N=1) | D150bid + ASA325qd (N=33) | D150qd + ASA325qd (N=1) | D300bid (N=105) | D300qd (N=3) | D300bid + ASA81qd (N=34) | D300qd + ASA81qd (N=2) | D300bid + ASA325qd (N=30) | D300qd + ASA325qd (N=1) | Warfarin (N=70)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2 | 3 | 3 | 0 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3 | 0 | 3 | 0 | 2 | 0 | 6 | 0 | 1 | 0 | 2 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 5 | 1 | 1 | 0 | 3
Sensation of pressure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 0 | 3 | 0 | 6
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 3 | 4 | 0 | 2 | 0 | 1 | 0 | 4 | 0 | 2 | 1 | 5 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 1 | 4 | 2 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 7 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 2 | 0 | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2
Exanthem (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.